CLINICAL TRIAL: NCT02517814
Title: Vitamin D Supplementation Can Improve Heart Function in Idiopathic Cardiomyopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HY-2015-06
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Cardiomyopathy, Dilated
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with cardiomyopathy (Experimental): Patients with vitamin D deficiency and cardiomyopathy will receive supplementation with vitamin D 400 units per day for 6 months.
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D

SUMMARY:
Vitamin D deficiency could be a high risk for cardiovascular diseases. It has been recently reported that vitamin D deficiency is another cause of heart failure and cardiomyopathies. It was found that vitamin D supplementation improved the heart function. The purpose of this study is to evaluate patients with idiopathic cardiomyopathies and determine whether vitamin D supplementation in cases where there is a deficiency, improves heart functioning.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic cardiomyopathy

Exclusion Criteria:

* Post heart surgery
* Congenital heart disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Improvement of heart function | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel